CLINICAL TRIAL: NCT01289054
Title: A Global Imatinib and Nilotinib Pregnancy Exposure Registry A Post-Authorisation Safety Study (PASS)
Brief Title: A Global Imatinib and Nilotinib Pregnancy Exposure Registry
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CSTI571A2403
Record Dates: First submitted 2011-01-31; First posted 2011-02-03 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: All Indications for Glivec/Gleevec and Tasigna
Keywords: Female; Pregnancy; Hematologic Pregnancy; Complications; Registry; Pregnant Registry; CML; GIST; Gleevec; Tasigna; Glivec; Pregnancy Exposure
MeSH Terms: interventions — nilotinib; Imatinib Mesylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort 1 - Pregnancy/Fetal Exposure
  Interventions: Drug: Tasigna; Drug: Gleevec
- Cohort 2 - Interrupted TKI

INTERVENTIONS:
Drug: Tasigna
  Groups: Cohort 1 - Pregnancy/Fetal Exposure
Drug: Gleevec
  Groups: Cohort 1 - Pregnancy/Fetal Exposure

SUMMARY:
This is a voluntary, international, primarily prospective, observational, exposure-registry and follow-up study of women receiving Imatinib and Nilotinib during pregnancy or within six months prior to pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Provide sufficient evidence to confirm that exposure occurred during pregnancy or within 6 months prior to exposure.
* Be at least 18 years of age
* Reside in a country supported by the Registry

Exclusion Criteria:

* Cases that do not meet the eligibility criteria are deemed ineligible, including paternal exposures

Other protocol-defined inclusion/exclusion criteria may apply

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women exposed to any dose of Gleevec/Glivec or Tasigna during pregnancy or within 6 months prior to conception
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Monitor pregnancies exposed to Imatinib or Nilotinib to estimate prevalence of birth defects | During pregnancy or within 6 months prior to conception

SECONDARY OUTCOMES:
Assess impact on maternal CML disease when treatment is interrupted | During pregnancy or within 6 months prior to conception
Assess post 12 month post-delivery data on maternal and infant status | 12 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- INC Research, LLC, Wilmington, North Carolina, United States